CLINICAL TRIAL: NCT02915835
Title: A Multi-center Randomized, Double Blind, Placebo-controlled, Pilot Study to Assess the Efficacy and Safety of Riociguat in Scleroderma - Associated Digital Ulcers
Brief Title: Riociguat in Scleroderma Associated Digital Ulcers
Acronym: RESCUE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Dinesh Khanna, MD, MS (Other)
Collaborators: Bayer (Industry)
Responsible Party: Sponsor-Investigator, Dinesh Khanna, MD, MS, Professor of Rheumatology/ Internal Medicine, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BAY63-2521
Record Dates: First submitted 2016-09-15; First posted 2016-09-27 (Estimated); Results first posted 2019-09-24 (Actual); Last update posted 2019-09-24 (Actual); Status verified 2019-09

CONDITIONS: Scleroderma; Digital Ulcers
Keywords: Scleroderma; Digital Ulcer
MeSH Terms: conditions — Scleroderma, Diffuse; digital ulcers | interventions — riociguat

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- riociguat (Active Comparator): Riociguat 0.5 mg, 1 mg, 1.5 mg, 2 mg and 2.5 mg administered TID; dose titration starting with 1.0 mg (planned up-titration every 2 weeks, with possibility of dose reduction for tolerability; 0.5 mg is the lowest dose and 2.5 mg is the highest dose to be administered)
  Interventions: Drug: Riociguat
- Placebo (Placebo Comparator): Matching placebo tablets: 0.5 mg, 1 mg, 1.5 mg, 2 mg and 2.5 mg administered TID; dose titration starting with 1.0 mg matching placebo tablet.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Riociguat — riociguat 0.5 mg, 1 mg, 1.5 mg, 2 mg and 2.5 mg administered TID; dose titration starting with 1.0 mg (planned up-titration every 2 weeks, with possibility of dose reduction for tolerability; 0.5 mg is the lowest dose and 2.5 mg is the highest dose to be administered)
  Other Names: Adempas
  Arms: riociguat
Drug: Placebo — Placebo 0.5 mg, 1 mg, 1.5 mg, 2 mg and 2.5 mg administered TID;
  Arms: Placebo

SUMMARY:
The primary objective of this study is to provide preliminary data on the efficacy (digital ulcer net burden) and safety of riociguat administered 3 times daily (TID) in comparison to placebo in patients with scleroderma-associated digital ulcers

DETAILED DESCRIPTION:
This clinical trial is a US, multicenter, double-blind, randomized placebo-controlled, parallel- group study with a total of 20 participants planned to be randomized (approximately 10 participants to the riociguat group and 10 to the placebo group). In addition, a standardized wound care protocol will be followed by the investigators and digital photography will be taken of the cardinal ulcer.

The study will allow standard of care medications for the management of DU as background therapy. These may include calcium channel blockers, low dose aspirin, angiotensin enzyme inhibitors, etc. and will be determined by the participant's local physician.

The study design consists of three phases:

* Screening phase: up to 2 weeks
* Double-blind Treatment phase: 16 weeks of double-blind treatment, consisting of:
* Dose titration period of up to 8 weeks, and
* Stable dosing period of up to 8 weeks
* Open-label Extension phase for participants with active DU at the end of the double- blind treatment phase or development of an active DU within a month of completing double-blind phase, consisting of:
* Dose titration phase of up to 8 weeks
* Stable dosing period for 8 weeks

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Men or women aged 18 years and older
3. Diagnosis of Systemic sclerosis, as defined by 2013 American College of Rheumatology/ European Union League Against Rheumatism classification of SSc
4. Patients had to have at least one visible, active ischemic DU at baseline located at or distal to the proximal interphalangeal joint, and that developed or worsened within 8 weeks prior to screening. NOTE: Presence of eschar will not be considered an active ulcer
5. Females of reproductive potential (FRP) must have a negative, pre-treatment urine pregnancy test.
6. FRP must obtain monthly urine pregnancy tests during treatment and one month after treatment discontinuation. Post-menopausal women (defined as no menses for at least 1 year or post-surgical from bilateral oophorectomy) are not required to undergo a pregnancy test.
7. FRP and all non-vasectomized male participants must agree to use reliable contraception when sexually active. (For FRP's, 'Adequate contraception' is defined as any combination of at least 2 effective methods of birth control, of which at least one is a physical barrier (e.g., condoms with hormonal contraception or implants or combined oral contraceptives, certain intrauterine devices). This applies from the time of signing the informed consent form until one month after the last study drug administration.)
8. Oral corticosteroids (≤ 10 mg/day of prednisone or equivalent), nonsteroidal anti- inflammatory drugs (NSAIDs), angiotensin receptor blockers, angiotensin converting enzyme (ACE) inhibitors and calcium channel blockers are permitted if the participant is on a stable dose for ≥ 2 weeks prior to and including the baseline visit
9. Ability to comply with the clinical visits schedule and the study-related procedures.

Exclusion Criteria:

1. Active DU related to calcinosis (as assessed by clinical examination or radiographic evaluation at screening)
2. Medical and surgical history

   * Major surgery (including joint surgery) within 8 weeks prior to screening
   * Participants with a history of malignancy in the last 5 years other than non-melanoma skin cell cancers cured by local resection or carcinoma in situ
3. Hepatic-related criteria

   - Hepatic insufficiency classified as Child-Pugh C at screening (see Appendix 11.1 for classification table) at screening visit
4. Renal-related criteria

   * Estimated glomerular filtration rate (eGFR) < 15 mL/min/1.73m2 (MDRD formula) or on dialysis at the screening visit
   * Cardiovascular-related criteria
   * Sitting systolic blood pressure < 95 mmHg at the screening visit
   * Sitting heart rate < 50 beats per minute (BPM) at the screening visit
   * Left ventricular ejection fraction < 40% prior to screening on echocardiogram done as part of clinical care
5. Pulmonary-related criteria

   * Active state of hemoptysis or pulmonary hemorrhage, including those events managed by bronchial artery embolization
   * Any history of bronchial artery embolization or massive hemoptysis within 3 months prior to screening. Massive hemoptysis being defined as acute bleeding >240 mL in a 24-hour period or recurrent bleeding >100 mL/d over several days
   * PAH requiring pharmacologic therapy.
   * Significant pulmonary disease with FVC ≤ 50% of predicted, or DLCO (uncorrected for hemoglobin ) ≤ 40% of predicted
6. Laboratory examinations

   - Participants with hemoglobin < 9.0 g/dL, white blood cell (WBC) count < 3000/mm3 (< 3 × 109/L), platelet count < 100,000/mm3 (< 3 × 109/L) at the screening visit
7. Prior and concomitant therapy

   * Concomitant use of nitrates or NO donors (such as amyl nitrate) in any form, including topical; phosphodiesterase (PDE) 5 (PDE5) inhibitors (such as sildenafil, tadalafil, vardenafil); and nonspecific PDE5 inhibitors (theophylline,dipyridamole). If the patient is on PDE5 inhibitors, a wash out of 3 days is required for sildenafil and 7 days for tadalafil or vardenafil prior to the baseline visit
   * Concomitant Endothelin receptor antagonist
   * Patients who are actively smoking at time of consent. (Quit date of two weeks prior to screening acceptable)
8. Pregnant or breastfeeding women
9. Other

   * Any other condition or therapy that would make the participant unsuitable for this study and will not allow participation for the full planned study period
   * Participation in another clinical study with an investigational drug or medical device within 30 days prior to randomization (phase I-III clinical studies)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2016-09; Primary Completion 2018-07-24 (Actual); Study Completion 2018-07-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dinesh Khanna, MD, Principal Investigator — University of Michigan
Locations (5):
- United States (5):
  - Georgetown University, Washington D.C., District of Columbia
  - University of Michigan, Ann Arbor, Michigan
  - Hospital of Special Surgery (HSS), New York, New York
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Nagaraja V, Spino C, Bush E, Tsou PS, Domsic RT, Lafyatis R, Frech T, Gordon JK, Steen VD, Khanna D. A multicenter randomized, double-blind, placebo-controlled pilot study to assess the efficacy and safety of riociguat in systemic sclerosis-associated digital ulcers. Arthritis Res Ther. 2019 Sep 3;21(1):202. doi: 10.1186/s13075-019-1979-7. PMID 31481106

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Riociguat | Placebo
Started | 9 | 8
Completed | 8 | 7
Not Completed | 1 | 1
Not completed — Physician Decision | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants who received at least one dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Riociguat | Placebo | Total
Number analyzed (Participants) | 9 | 8 | 17
Age, Continuous [Mean (Standard Deviation); unit: years] | 43 (14) | 61 (17) | 51 (18)
Age, Customized [Count of Participants; unit: Participants]
  Age Categories: 18 to 35 years | 4 | 1 | 5
  Age Categories: >35 to 55 years | 3 | 1 | 4
  Age Categories: >55 to 75 years | 2 | 5 | 7
  Age Categories: >75 years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 5 | 13
  Male | 1 | 3 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 8 | 17
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 6 | 7 | 13
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Number of digital ulcers at screening [Mean (Standard Deviation); unit: number of digital ulcers] — defined as active and painful indeterminate digital ulcers
  number of digital ulcers | 2.67 (1.803) | 2.50 (1.690) | 2.59 (1.698)
Type of scleroderma at screening [Count of Participants; unit: Participants]
  limited cutaneous | 5 | 4 | 9
  diffuse cutaneous | 4 | 4 | 8
Time since first non-Raynaud's Symptom [Mean (Standard Deviation); unit: years] — time since first non-Raynaud's symptom until screening visit
  years | 7.09 (5.933) | 17.49 (11.09) | 11.98 (10.060)
Time since first Raynaud's Phenomenon symptom [Mean (Standard Deviation); unit: years] — Time since first Raynaud's Phenomenon symptom until the screening visit
  years | 7.49 (6.649) | 14.5 (7.872) | 11.01 (7.920)
Time since Scleroderma Diagnosis [Mean (Standard Deviation); unit: years] — Time since the diagnosis of scleroderma until the screening visit
  years | 6.23 (5.765) | 15.0 (8.05) | 10.37 (8.156)
Time since first Digital Ulcer [Mean (Standard Deviation); unit: years] | 5.41 (4.563) | 8.07 (6.842) | 6.66 (5.725)
SHAQ: Finger ulcers interfere with daily activities in past week [Median (Inter-Quartile Range); unit: units on a scale] — The Scleroderma Health Assessment Questionnaire (SHAQ) visual analogue scale assessing the burden of digital ulcers (In the past week, how much have your finger ulcers interfered with your daily activities?). The score indicates degree of limitation of activity from a scale of 0 (no limitation) to 150 (most limitation).
  units on a scale | 116 [98 to 125] | 55 [36 to 102] | 98 [62 to 124]
Raynaud's condition score [Mean (Standard Deviation); unit: units on a scale] — The Raynaud's condition score is a daily patient assessment of Raynaud's phenomenon activity using a 0 -10 ordinal scale. It incorporates the cumulative frequency, duration, severity and impact of Raynaud's phenomenon attacks, reflecting the overall degree that Raynaud's has affected use of the participant's hands. A score of 0 indicates no difficulty and 10 indicates extreme difficulty with Raynaud's condition.
  units on a scale | 3.4 (2.2) | 5.4 (1.6) | 4.5 (2.1)
Number of Raynaud's attacks per day [Mean (Standard Deviation); unit: attacks per day] — The number of Raynaud's attacks is the mean number of Raynaud's attacks per day over a 7-day period.
  attacks per day | 4.3 (1.7) | 2.2 (1.7) | 3.3 (2.0)
Pain during a Raynaud's attack [Mean (Standard Deviation); unit: units on a scale] — Pain because of Raynaud's disease (characterized as pain during a Raynaud's attack) is defined on a visual analogue scale, where 0 indicates no pain and 100 indicates very severe pain. The mean of the scales over a 7-day period are reported.
  units on a scale | 54.9 (13.1) | 37.2 (24.6) | 46.6 (20.7)
Numbness during a Raynaud's attack [Mean (Standard Deviation); unit: units on a scale] — Numbness because of Raynaud's disease (characterized as numbness during a Raynaud's attack) is defined on a visual analogue scale, where 0 indicates no numbness and 100 indicates very severe numbness. The mean of the scales over a 7-day period are reported.
  units on a scale | 40.5 (15.9) | 32.0 (30.2) | 36.5 (23.2)
Tingling during a Raynaud's attack [Mean (Standard Deviation); unit: units on a scale] — Tingling because of Raynaud's disease (characterized as tingling during a Raynaud's attack) is defined on a visual analogue scale, where 0 indicates no tingling and 100 indicates very severe tingling. The mean of the scales over a 7-day period are reported.
  units on a scale | 34.8 (16.6) | 26.9 (16.1) | 31.1 (16.3)
Duration of Raynaud's attacks [Mean (Standard Deviation); unit: minutes] — The mean duration of a Raynaud's attack (in minutes) is calculated across a 7-day period. For the days when a participant does not have an attack, a value of 0 is used in the calculation.
  minutes | 101.4 (117.3) | 47.9 (51.6) | 76.4 (93.8)
Severity of patient assessment of Raynaud's phenomenon [Mean (Standard Deviation); unit: units on a scale] — The severity of Raynaud's phenomenon, as assessed by the patient, ranges from 0 (not at all severe) to 10 (extremely severe).
  units on a scale | 7.1 (1.4) | 4.2 (2.7) | 5.8 (2.5)
Severity of patient assessment of digital ulcers [Mean (Standard Deviation); unit: units on a scale] — The severity of digital ulcers, as assessed by the patient, ranges from 0 (not at all severe) to 10 (extremely severe).
  units on a scale | 8.0 (1.5) | 6.7 (1.9) | 7.4 (1.8)
Severity of physician assessment of Raynaud's phenomenon [Mean (Standard Deviation); unit: units on a scale] — The severity of Raynaud's phenomenon, as assessed by the physician, ranges from 0 (not at all severe) to 10 (extremely severe).
  units on a scale | 6.1 (1.0) | 5.4 (3.0) | 5.8 (2.1)
Severity of physician assessment of digital ulcers [Mean (Standard Deviation); unit: units on a scale] — The severity of digital ulcers, as assessed by the physician, ranges from 0 (not at all severe) to 10 (extremely severe).
  units on a scale | 6.4 (1.9) | 6.3 (2.6) | 6.4 (2.1)
Systemic scleroderma-related antibodies [Count of Participants; unit: Participants]
  Anti-centromere B | 3 | 3 | 6
  Anti-topoisomerase I | 2 | 3 | 5
  Anti-RNA polymerase III | 1 | 0 | 1
  Not done | 3 | 2 | 5
Baseline use of vasodilators [Count of Participants; unit: Participants] | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to End of Double-blind Treatment (Week 16) in Digital Ulcer Net Burden
Description: Digital ulcer net burden is defined as the total number of "active" and indeterminate digital ulcers at an assessment. Active ulcers are defined as having a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity. A healed ulcer has complete re-epithelialization.
Time Frame: Baseline to Week 16
Population: Modified Intent to Treat Population is defined as all participants randomized, receiving at least one dose of treatment, and having at least one post-baseline efficacy assessment.
Measure: Least Squares Mean (Standard Error); unit: ulcers
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
ulcers | -1.22 (0.458) | -0.98 (0.425)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.70, ANCOVA

2. Secondary Outcome: Proportion of Participants With Healing of Their Cardinal DU by Week 16
Description: The proportion of participant whose active digital ulcer that was identified and designated by the investigator as the cardinal ulcer at Baseline is healed by week 16. The cardinal ulcer will be selected by the investigator based on the clinical judgment that it was amenable to and evaluable for healing. If there are several active digital ulcers, the cardinal ulcer could be either the largest or the most painful ulcer, or the ulcer that disturbed the patient the most. Active ulcers are defined as having a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis.
Time Frame: Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 4 | 6
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.61, Fisher Exact

3. Secondary Outcome: Proportion of Participants With Healing of All DUs at Baseline by Week 16
Description: The proportion of participants whose baseline DUs are considered healed (classified as 'healed' and not 'active' or 'indeterminate') by week 16. All baseline ulcers must be healed for the participant to be classified as having all baseline ulcers healed. Note that this end point does not consider whether a participant develops new DUs during the course of the study. Active ulcers are defined as having a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity. A healed ulcer has complete re-epithelialization.
Time Frame: Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 3 | 3
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

4. Secondary Outcome: Proportion of Participants With no DUs at Week 16
Description: The proportion of participants with no digital ulcers at week 16. This end point does not consider the number of ulcers at baseline or during the course of the study; only the absence of 'active' and 'indeterminate' DUs at week 16. Active ulcers are defined as having a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity. A healed ulcer has complete re-epithelialization.
Time Frame: Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 2 | 2
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

5. Secondary Outcome: Proportion of Participants With New Active and Indeterminate DU(s) Over the Course of the Double-blind Period
Description: The proportion of participants with new (i.e., not present at baseline) active and indeterminant DUs from baseline to Week 16. An active ulcer is defined as a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 3 | 4
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

6. Secondary Outcome: Proportion of Participants Who Develop Pressure Ulcers at Distal Interphalangeal (DIP) Location Over the Course of the Double-blind Period.
Description: The proportion of participants who develop a DIP pressure ulcer at baseline to Week 16. Pressure ulcer is defined as an active or indeterminate ulcer. An active ulcer is defined as a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 0 | 1
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

7. Secondary Outcome: Proportion of Participants Who Develop Pressure Ulcers at Proximal Interphalangeal (PIP) Location Over the Course of the Double-blind Period.
Description: The proportion of participants who develop a PIP pressure ulcer at baseline to Week 16. Pressure ulcer is defined as an active or indeterminate ulcer. An active ulcer is defined as a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 1 | 2
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

8. Secondary Outcome: Proportion of Participants Who Develop Pressure Ulcers at Metacarpophalangeal (MCPs) Location Over the Course of the Double-blind Period.
Description: The proportion of participants who develop a MCP pressure ulcer at baseline to Week 16. Pressure ulcer is defined as an active or indeterminate ulcer. An active ulcer is defined as a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

9. Secondary Outcome: Proportion of Participants Who Develop Pressure Ulcers at the Elbows Over the Course of the Double-blind Period.
Description: The proportion of participants who develop a pressure ulcer at at the elbows at baseline to Week 16. Pressure ulcer is defined as an active or indeterminate ulcer. An active ulcer is defined as a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

10. Secondary Outcome: Proportion of Participants With Healing of All Pressure Ulcers at the Distal Interphalangeal (DIP) Over the Course of the Double-blind Period.
Description: The proportion of participants whose DIP pressure ulcers during the double-blind period were healed at Week 16. Pressure ulcer is defined as an active or indeterminate ulcer. An active ulcer is defined as a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

11. Secondary Outcome: Proportion of Participants With Healing of All Pressure Ulcers at the Proximal Interphalangeal (PIP) Over the Course of the Double-blind Period.
Description: The proportion of participants whose PIP pressure ulcers during the double-blind period were healed at Week 16. Pressure ulcer is defined as an active or indeterminate ulcer. An active ulcer is defined as a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 1 | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

12. Secondary Outcome: Proportion of Participants With Healing of All Pressure Ulcers at the Metacarpophalangeal (MCPs) Over the Course of the Double-blind Period.
Description: The proportion of participants whose MCP pressure ulcers during the double-blind period were healed at Week 16. Pressure ulcer is defined as an active or indeterminate ulcer. An active ulcer is defined as a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

13. Secondary Outcome: Proportion of Participants With Healing of All Pressure Ulcers at the Elbows Over the Course of the Double-blind Period.
Description: The proportion of participants whose pressure ulcers at the elbows during the double-blind period were healed at Week 16. Pressure ulcer is defined as an active or indeterminate ulcer. An active ulcer is defined as a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 8 | 8
Participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

14. Secondary Outcome: Time to Healing of Cardinal DU
Description: This is defined as the number of weeks from randomization to the earliest of healing, end of the double-blind period, or drop-out. Participants are censored if they drop-out or their cardinal DU has not healed by the end of the double-blind period. One active digital ulcer must be identified and designated by the investigator as the cardinal ulcer at Baseline. If several digital ulcers qualified, the cardinal ulcer could be either the largest or the most painful ulcer, or the ulcer that disturbed the patient the most. The cardinal ulcer will be selected by the investigator based on the clinical judgment that it was amenable to and evaluable for healing. Active ulcers are defined as having a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. Week 16 is defined as the end of the double-blind period; however, the protocol allowed a visit window of +/- 4 weeks.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
weeks | 16.57 [2.00 to 17.57] | 16.07 [16.00 to 16.14]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .56, Log Rank

15. Secondary Outcome: Time to Healing of All Baseline DU
Description: This is defined as the number of weeks from randomization to the earliest of all baseline DU(s) healed, end of the double-blind period, or drop-out. Participants are censored if they drop-out or all of their baseline DU(s) have not healed by the end of the double-blind period. A healed ulcer has complete re-epithelialization. Week 16 is defined as the end of the double-blind period; however, the protocol allowed a visit window of +/- 4 weeks.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
weeks | 16.00 [2.00 to 16.86] | 16.00 [14.86 to 16.43]
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .35, Log Rank

16. Secondary Outcome: Time to Development of New ('Active' or 'Indeterminate') DU
Description: This is defined as the number of weeks from randomization to the earliest of new DU, end of the double-blind period, or drop-out. Participants are censored if they drop-out or have not developed a new DU by the end of the double-blind period. Active ulcers are defined as having a denuded area with defined border and loss of epithelialization, loss of epidermis and dermis. An indeterminate ulcer is defined as denudation that could not be visualized and no other clinical features of activity. A healed ulcer has complete re-epithelialization. Week 16 is defined as the end of the double-blind period; however, the protocol allowed a visit window of +/- 4 weeks.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
weeks | 16.00 [15.71 to 16.86] | 15.86 [15.57 to 16.43]

17. Secondary Outcome: Change From Baseline to Week 16 in Raynaud's Condition Score
Description: The Raynaud's condition score is a daily patient assessment of Raynaud's phenomenon activity using a 0 -10 ordinal scale. It incorporates the cumulative frequency, duration, severity and impact of Raynaud's phenomenon attacks, reflecting the overall degree that Raynaud's has affected use of the participant's hands. A score of 0 indicates no difficulty and 10 indicates extreme difficulty with Raynaud's condition. A higher score means a worse outcome. The mean score will be calculated across the 7-day screening and week 16 periods for each participant.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -1.15 (.691) | -0.82 (.691)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .76, ANCOVA

18. Secondary Outcome: Change From Baseline to Week 16 in Number of Raynaud's Attacks/Day
Description: The mean number of Raynaud's attacks each day will be calculated across the 7-day screening and week 16 periods for each participant. For the days when a participant does not have an attack, a score of 0 will be used.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: attacks per day
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
attacks per day | -1.24 (.323) | -0.96 (.323)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .57, ANCOVA

19. Secondary Outcome: Change From Baseline to Week 16 in Duration of Raynaud's Attacks
Description: The mean duration of attacks (in minutes) will be calculated across the 7-day screening and week 16 periods for each participant. For the days when a participant does not have an attack, a score of 0 will be used.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
minutes | -44.81 (15.846) | 150.3 (15.846)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .40, ANCOVA

20. Secondary Outcome: Change From Baseline to Week 16 in Patient's Assessment of Pain During a Raynaud's Attack
Description: Pain because of Raynaud's disease (characterized as pain during a Raynaud's attack) is defined on a visual analogue scale, where 0 indicates no pain and 100 indicates very severe pain. A higher score means a worse outcome. The mean of the scales over a 7-day period are reported. For the days when a participant does not have an attack, a score of 0 will be used. The mean scale score for each symptom will be calculated across the 7-day screening and week 16 periods for each participant.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -0.30 (6.600) | -7.01 (6.600)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .49, ANCOVA

21. Secondary Outcome: Change From Baseline to Week 16 in Patient's Assessment of Numbness During a Raynaud's Attack
Description: Numbness because of Raynaud's disease (characterized as numbness during a Raynaud's attack) is defined on a visual analogue scale, where 0 indicates no numbness and 100 indicates very severe numbness. A higher score means a worse outcome. The mean of the scales over a 7-day period are reported. For the days when a participant does not have an attack, a score of 0 will be used. The mean scale score for each symptom will be calculated across the 7-day screening and week 16 periods for each participant.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -19.73 (8.899) | -15.44 (8.899)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .75, ANCOVA

22. Secondary Outcome: Change From Baseline to Week 16 in Patient's Assessment of Tingling During a Raynaud's Attack
Description: Tingling because of Raynaud's disease (characterized as tingling during a Raynaud's attack) is defined on a visual analogue scale, where 0 indicates no tingling and 100 indicates very severe tingling. A higher score means a worse outcome. The mean of the scales over a 7-day period are reported. For the days when a participant does not have an attack, a score of 0 will be used. The mean scale score for each symptom will be calculated across the 7-day screening and week 16 periods for each participant.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | 1.18 (7.118) | -7.49 (7.118)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .41, ANCOVA

23. Secondary Outcome: Change From Baseline to Week 16 in Physician's Assessment of Severity of Raynaud's Disease
Description: The severity of Raynaud's phenomenon, as assessed by the physician, ranges from 0 (not at all severe) to 10 (extremely severe). A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -3.00 (0.736) | -1.86 (0.788)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.31, ANCOVA

24. Secondary Outcome: Change From Baseline to Week 16 in Physician's Assessment of Severity of Digital Ulcers
Description: The severity of digital ulcers, as assessed by the physician, ranges from 0 (not at all severe) to 10 (extremely severe). A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -3.54 (0.886) | -3.81 (0.948)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.84, ANCOVA

25. Secondary Outcome: Change From Baseline to Week 16 in Patient's Assessment of Severity of Raynaud's Disease
Description: The severity of Raynaud's phenomenon, as assessed by the patient, ranges from 0 (not at all severe) to 10 (extremely severe). A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: Severity of Raynaud's disease is calculated as the mean response on a 0-10 Likert scale.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -3.47 (0.764) | -1.41 (0.764)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.11, ANCOVA

26. Secondary Outcome: Change From Baseline to Week 16 in Patient's Assessment of Severity of Digital Ulcers
Description: The severity of digital ulcers, as assessed by the patient, ranges from 0 (not at all severe) to 10 (extremely severe). A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: Severity of digital ulcer(s) is calculated as the mean response on a 0-10 Likert scale.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -4.63 (0.935) | -4.00 (0.935)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.66, ANCOVA

27. Secondary Outcome: Change From Baseline to Week 16 in Patient's Global Assessment for Overall Disease.
Description: This assessment represents the patient's assessment of the patient's global scleroderma on a 0 (excellent) -10 (extremely poor) Likert scale. A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | 0.31 (0.915) | -1.19 (0.915)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.27, ANCOVA

28. Secondary Outcome: Change From Baseline to Week 16 in Physician's Global Assessment for Overall Disease.
Description: This assessment represents the physician's assessment of the patient's current disease activity on a 0 (excellent) -10 (extremely poor) Likert scale. A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
units on a scale | -1.17 (0.548) | -0.66 (0.586)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.54, ANCOVA

29. Secondary Outcome: Change From Baseline to Week 16 in PROMIS-29 Physical Function
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the physical function domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., better outcome).
Time Frame: Baseline/Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
t-score | -2.46 (1.27) | -2.24 (1.227)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .90, ANCOVA

30. Secondary Outcome: Change From Baseline to Week 16 in PROMIS-29 Anxiety
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the anxiety domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).y.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
t-score | -3.11 (2.578) | -1.50 (2.578)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .68, ANCOVA

31. Secondary Outcome: Change From Baseline to Week 16 in PROMIS-29 Depression
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the depression domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
t-score | -3.35 (1.731) | -0.25 (1.731)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .25, ANCOVA

32. Secondary Outcome: Change From Baseline to Week 16 in PROMIS-29 Fatigue
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the fatigue domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
t-score | 0.64 (1.903) | 0.46 (1.903)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .95, ANCOVA

33. Secondary Outcome: Change From Baseline to Week 16 in PROMIS-29 Sleep Disturbance
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the sleep disturbance domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e.,worse outcome).
Time Frame: Baseline/Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
t-score | -0.47 (1.091) | 0.94 (1.091)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.38, ANCOVA

34. Secondary Outcome: Change From Baseline to Week 16 in PROMIS-29 Pain Interference
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the pain interference domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
t-score | -3.69 (1.798) | -3.06 (1.798)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .82, ANCOVA

35. Secondary Outcome: Change From Baseline to Week 16 in PROMIS-29 Ability to Participate in Social Roles and Activities
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the ability to participate in social roles and activities domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., better outcome).
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
t-score | -1.68 (1.104) | -0.46 (1.104)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = .47, ANCOVA

36. Secondary Outcome: Change From Baseline to Week 16 in PROMIS-29 Pain Intensity
Description: The Patient-Reported Outcomes Measurement Information System (PROMIS) 29-item short-form health-reported quality of life measures (PROMIS-29) were administered. The transformed score (T-score) for the pain intensity domain was used, where 50 (10) is the mean (standard deviation) of a relevant reference population. Higher scores equals more of the concept being measured (i.e., worse outcome).
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: t-score
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
t-score | -2.74 (0.702) | -1.63 (0.702)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.35, ANCOVA

37. Secondary Outcome: Change From Baseline to Week 16 in Overall HAQ-DI Score
Description: The HAQ-DI is the Health Assessment Question Disability Index that assesses the extent of a patient's functional ability. The HAQ-DI overall score ranges from 0 (no disability) to 3 (severe disability). Higher score means worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -0.01 (0.149) | -0.06 (0.160)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.84, ANCOVA

38. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI Dressing and Grooming
Description: The HAQ-DI is the Health Assessment Question Disability Index that assesses the extent of a patient's functional ability. The HAQ-DI subscore ranges from 0 (no disability) to 3 (severe disability). A higher score means worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -0.16 (0.18) | 0.05 (0.236)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.55, ANCOVA

39. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI Hygiene
Description: as for outcome 38
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -0.39 (0.279) | -0.27 (0.298)

40. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI Arising
Description: as for outcome 38
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | 0.36 (0.235) | 0.02 (0.251)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.34, ANCOVA

41. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI Reach
Description: as for outcome 38
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | 0.37 (0.253) | 0.01 (0.271)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.36, ANCOVA

42. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI Eating
Description: as for outcome 38
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -0.53 (0.154) | 0.03 (0.166)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.04, ANCOVA

43. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI Grip
Description: as for outcome 38
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | 0.16 (0.215) | -0.18 (0.230)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.32, ANCOVA

44. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI Walking
Description: as for outcome 38
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | 0.35 (0.199) | -0.12 (0.214)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.14, ANCOVA

45. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI Common Daily Activities (IADL).
Description: as for outcome 38
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -0.29 (0.260) | 0.04 (0.278)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.41, ANCOVA

46. Secondary Outcome: Change From Baseline to Week 16 in HAQ-DI Composite Score for Hand Function
Description: The HAQ-DI is the Health Assessment Question Disability Index that assesses the extent of a patient's functional ability. The HAQ-DI subscore ranges from 0 (no disability) to 3 (severe disability).The sum of the individual scores for dressing, hygiene, and grip from the HAQ-DI defines the composite score for hand function. The HAQ-DI composite score for hand function ranges from 0 (no disability) to 9 (severe disability). A higher score means worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -0.47 (0.492) | -0.32 (0.527)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.85, ANCOVA

47. Secondary Outcome: Change From Baseline to Week 16 in Total Hand Disability in Systemic Sclerosis-DU (HDISS-DU) Score
Description: The Hand Disability in Systemic Sclerosis - Digital Ulcers (HDISS-DU) questionnaire is a 24-item PRO measure. Each item is scored from 1-6 (1=yes, without difficulty; 2=yes, with a little difficulty; 3=yes, with some difficulty; 4=yes with much difficulty; 5=nearly impossible to do & used unaffected hand only; 6=impossible). The total HDISS-DU score is the mean of valid items, ranging from 1 to 6. Higher scores represent increased disability in hand functioning.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -0.47 (0.492) | -0.32 (0.527)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.85, ANCOVA

48. Secondary Outcome: Change From Baseline to Week 16 in Scleroderma-HAQ-DI Visual Analogue Scales (VAS) Assessing Burden of Digital Ulcers
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for how much finger ulcers interfered with daily activities ranges from 0 (do not limit activities) to 150 (very severe limitation). A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -43.09 (18.457) | -53.47 (20.159)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.75, ANCOVA

49. Secondary Outcome: Change From Baseline to Week 16 in Scleroderma-HAQ-DI Visual Analogue Scales (VAS) Assessing Raynaud's Disease
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for how much Raynaud's interfered with daily activities ranges from 0 (does not limit activities) to 150 (very severe limitation). A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -23.78 (15.6) | -25.40 (16.982)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.95, ANCOVA

50. Secondary Outcome: Change From Baseline to Week 16 in Scleroderma-HAQ-DI Visual Analogue Scales (VAS) Assessing Gastrointestinal Involvement
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for how much intestinal problems interfered with daily activities ranges from 0 (do not limit activities) to 150 (very severe limitation). A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | 16.72 (13.787) | -7.39 (14.975)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.31, ANCOVA

51. Secondary Outcome: Change From Baseline to Week 16 in Scleroderma-HAQ-DI Visual Analogue Scales (VAS) Assessing Breathing
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for how much breathing problems interfered with daily activities ranges from 0 (do not limit activities) to 150 (very severe limitation). A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | 8.35 (8.90) | -12.69 (8.978)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.14, ANCOVA

52. Secondary Outcome: Change From Baseline to Week 16 in Scleroderma-HAQ-DI Visual Analogue Scales (VAS) Assessing Overall Disease,
Description: Scleroderma-Health Assessment Question Disability Index visual analogue scales (VAS) assess the burden of digital ulcers, Raynaud's, gastrointestinal involvement, breathing, and overall disease. The VAS scale for disease severity ranges from 0 (no disease) to 150 (very severe). A higher score means a worse outcome.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
score on a scale | -50.35 (9.039) | -35.74 (9.751)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.32, ANCOVA

53. Secondary Outcome: Proportion of Participants Who Experience Digital Ischemia Requiring Intravenous Prostacyclin or Digital Gangrene or Amputation During the Trial.
Description: The proportion of participants who experience digital ischemia requiring intravenous prostacyclin or digital gangrene or amputation during the double-blind period of the trial. These outcomes are collected within Adverse Events
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
Participants | 0 | 1
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.47, Fisher Exact

54. Secondary Outcome: Proportion of Participants Who Develop Osteomyelitis During The Trial
Description: The proportion of participants who developed osteomyelitis during the double-blind period of the trial. Osteomyelitis is collected as an Adverse Event.
Time Frame: Baseline to Week 16
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
Participants | 0 | 0
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 1.00, Fisher Exact

55. Secondary Outcome: Change From Baseline to Week 16 in Vascular Biomarker VEGF in the Plasma
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
pg/ml | -29.8 (9.5) | -34.7 (10.1)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.73, ANCOVA

56. Secondary Outcome: Change From Baseline to Week 16 in Vascular Biomarker tPA in the Plasma
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
ng/ml | -1.2 (0.5) | -0.5 (0.5)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.32, ANCOVA

57. Secondary Outcome: Change From Baseline to Week 16 in Vascular Biomarker sE-Selectin in the Plasma
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
ng/ml | -4.7 (1.9) | -2.5 (2.0)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.45, ANCOVA

58. Secondary Outcome: Change From Baseline to Week 16 in Vascular Biomarker BFGF in the Plasma
Time Frame: Baseline and Week 16
Measure: Least Squares Mean (Standard Error); unit: pg/ml
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
pg/ml | 0.20 (0.28) | -0.03 (0.29)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.58, ANCOVA

59. Secondary Outcome: Change From Baseline to Week 16 in Vascular Biomarker VCAM-1 in the Plasma
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
ng/ml | 10.3 (10.4) | -3.4 (11.0)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.39, ANCOVA

60. Secondary Outcome: Change From Baseline to Week 16 in Vascular Biomarker ICAM in the Plasma
Time Frame: Baseline and Week 16
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: ng/ml
Arm/Group | Riociguat | Placebo
Number analyzed (Participants) | 9 | 8
ng/ml | 70.5 (47.3) | -39. (50.2)
Statistical Analysis 1: Comparison: Placebo; Test type: Superiority; p = 0.14, ANCOVA

ADVERSE EVENTS:
Time Frame: 16 weeks
Description: Coding of adverse events into body system was performed by the study chair for adverse events and by the medical monitors for serious adverse events.
Arm/Group | Riociguat | Placebo
All-Cause Mortality (participants affected / at risk) | 0/9 | 0/8
Serious Adverse Events (participants affected / at risk) | 3/9 | 1/8
Other Adverse Events (participants affected / at risk) | 9/9 | 8/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (N=9) | Placebo (N=8)
Lymphoma (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
NSTEMI (Cardiac disorders) | 1 (1) | 0 (0)
Digital ischemia of the right third toe (Vascular disorders) | 0 (0) | 1 (1)
Right 4th digit ulcer (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Riociguat (N=9) | Placebo (N=8)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Splenic infarct (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Heart Murmur (Cardiac disorders) | 1 (1) | 0 (0)
Left bundle bramch block on EKG (Cardiac disorders) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 1 (1)
GERD (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Hot flashes (General disorders) | 0 (0) | 1 (1)
Elevated liver enzymes (Hepatobiliary disorders) | 1 (1) | 0 (0)
Right calf infection (Infections and infestations) | 0 (0) | 1 (1)
Ulcer infection (Infections and infestations) | 2 (2) | 0 (0)
Right arm laceration (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Calcinosis Ulcer over Right Knee (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left Shoulder Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Left Shoulder rotator cuff tear (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Left elbow bursitis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 3 (3) | 3 (3)
Lightheadednes (Nervous system disorders) | 2 (2) | 1 (1)
Shoulder surgery (Surgical and medical procedures) | 0 (0) | 1 (1)
Cyanosis (Vascular disorders) | 0 (0) | 1 (1)
Worsening Raynaud's (Vascular disorders) | 1 (1) | 0 (0)
Worsening digital ulcer (Vascular disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/35/NCT02915835/Prot_000.pdf
  • Statistical Analysis Plan (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/35/NCT02915835/SAP_001.pdf